CLINICAL TRIAL: NCT03896477
Title: A Phase 3, Randomized, Observer-Blind Study to Evaluate the Safety, Tolerability, Immunogenicity of Serum Institute of India's 10-Valent Pneumococcal Conjugate Vaccine (PNEUMOSIL®) Administered in a 2+1 Schedule to Healthy Infants in The Gambia
Brief Title: Study of 10-valent Pneumococcal Conjugate Vaccine (Pneumosil) Administered in a 2+1 Schedule to Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Serum Institute of India Pvt. Ltd. (Industry); Medical Research Council Unit, The Gambia (Other); University College, London (Other); FHI 360 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CVIA-074; PACTR201907754270299 (Registry Identifier: Pan African Clinical Trials Registry)
Record Dates: First submitted 2019-03-22; First posted 2019-04-01 (Actual); Results first posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumococcal
MeSH Terms: conditions — Pneumonia, Pneumococcal | interventions — 13-valent pneumococcal vaccine; PHiD-CV vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pneumosil (Experimental): Infants received two primary vaccinations with Pneumosil, the first at age 6 weeks and the second at age 14 weeks. A booster vaccination was given between 9 and 16 months of age.
  Interventions: Biological: Pneumosil
- Synflorix (Active Comparator): Infants received two primary vaccinations with Synflorix, the first at age 6 weeks and the second at age 14 weeks. A booster vaccination was given between 9 and 16 months of age.
  Interventions: Biological: Synflorix
- Prevenar 13 (Active Comparator): Infants received two primary vaccinations with Prevenar 13, the first at age 6 weeks and the second at age 14 weeks. A booster vaccination was given between 9 and 16 months of age.
  Interventions: Biological: Prevenar 13

INTERVENTIONS:
Biological: Pneumosil — One single dose contains 2 μg of polysaccharide for serotypes 1, 5, 6A, 7F, 9V, 14, 19A, 19F and 23F, and 4 μg for serotype 6B formulated with aluminium phosphate as an adjuvant in an appropriate buffer
  Other Names: Serum Institute of India Pneumococcal conjugate vaccine (SIIPL-PCV )
  Arms: Pneumosil
Biological: Prevenar 13 — One single dose contains 2.2 µg of the following pneumococcal polysaccharides serotypes - 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F - and 4.4 µg of pneumococcal polysaccharide serotype 6B, all conjugated to CRM197 and absorbed onto aluminum phosphate
  Arms: Prevenar 13
Biological: Synflorix — One single dose contains 1 μg of polysaccharide for serotypes 1, 5, 6B, 7F, 9V, 14, and 23F, and 3μg of serotypes 4, 18C, and 19F formulated with aluminum phosphate as an adjuvant.
  Other Names: Pneumococcal polysaccharide conjugate vaccine (adsorbed)
  Arms: Synflorix

SUMMARY:
The primary objectives of this study are to evaluate the immunogenicity (antibody response) and safety and tolerability of a 2-dose primary series and booster dose (2+1 schedule) of Pneumosil co-administered with routine pediatric vaccines in healthy infants in The Gambia.

DETAILED DESCRIPTION:
This study will provide data necessary to evaluate the safety and immunogenicity of Pneumosil when administered in an alternative schedule to the 3 dose primary schedule (3+0) evaluated in the Phase 3 pivotal trial (VAC-056; NCT03197376) - namely in a 2 dose primary and booster (2+1) schedule - and compare immunogenicity to that of both currently licensed second-generation pneumococcal conjugate vaccines (Synflorix and Prevenar 13) administered in the same 2+1 schedule.

In this prospective, single center, randomized, active-controlled, observer-blind, Phase 3 descriptive study, 660 healthy Gambian pneumococcal conjugate vaccine (PCV)-naïve infants will be randomized 1:1:1 to receive 3 doses of either Pneumosil, Synflorix or Prevenar 13 at 6 weeks, 14 weeks and 9-10 months of age. Standard Expanded Program on Immunization (EPI) vaccinations in The Gambia will be given concomitantly with all 3 doses of study vaccine.

The booster vaccination window was extended up to 18 months of age due to a pause in the study due to the coronavirus disease 2019 (COVID-19) pandemic. The study schedule for participants is as follows:

* Age 6 weeks: First primary vaccination dose administered
* Age 14 weeks: Second primary vaccination dose administered (8 weeks after first primary dose)
* Age 18 weeks: Blood sample for immunogenicity testing (4 weeks after second primary dose)
* Age 9-18 months: Blood sample for immunogenicity testing and booster vaccination dose administered
* Age 10-19 months: Blood sample for immunogenicity testing (4 weeks after booster dose)

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants based on medical history and clinical assessment.
* Between 6 and 8 weeks (ie 42 to 56 days) old, inclusive.
* Subject's parent must provide voluntary written/thumb-printed informed consent and be willing to comply with study requirements and procedures.
* Subjects must have been born full-term, have a weight-to-height Z score of ≥ -2 at the time of enrollment (WHO child growth standard), and be ≥ 3.5 kg at randomization.
* Subject's parents must be available for the duration of trial participation

Exclusion Criteria:

* Use of any investigational medicinal product prior to randomization.
* Previous vaccination against or infection with S. pneumoniae.
* History of anaphylactic shock or an allergic reaction to any prior vaccination.
* Any fever, illness (including malaria).
* Receipt of another study vaccine within 30 days of study start.
* Chronic administration of an immunosuppressant or administration of immunoglobulins
* History of blood disorder, primary immunodeficiency, or a sibling who has such a diagnosis or who died suddenly without apparent cause.
* History of meningitis, seizures or any neurological disorder.
* Exposure to human immunodeficiency virus (HIV) by history.

Ages: 42 Days to 56 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 660 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ed Clarke, MB ChB, PhD, Principal Investigator — MRCG at LSHTM
Locations (1):
- Medical Research Council Unit, The Gambia at the London School of Hygiene and Tropical Medicine (MRCG at LSHTM), Banjul, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adigweme I, Futa A, Saidy-Jah E, Edem B, Akpalu E, Dibbasey T, Sethna V, Dhere R, Kampmann B, Bengt C, Sirr J, Hosken N, Goldblatt D, Antony K, Alderson MR, Lamola S, Clarke E. Immunogenicity and safety of a 10-valent pneumococcal conjugate vaccine administered as a 2 + 1 schedule to healthy infants in The Gambia: a single-centre, double-blind, active-controlled, randomised, phase 3 trial. Lancet Infect Dis. 2023 May;23(5):609-620. doi: 10.1016/S1473-3099(22)00734-4. Epub 2023 Jan 10. PMID 36638819

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy, Gambian male and female, pneumococcal conjugate vaccine (PCV)-naïve infants were screened and enrolled at the Medical Research Council Unit, The Gambia at the London School of Hygiene and Tropical Medicine (MRCG at LSHTM).
Pre-assignment Details: Eligible participants were randomized equally (in a 1:1:1 ratio), based on a pre-established randomization scheme, to receive either Pneumosil, Synflorix or Prevenar 13. Participants were to receive two primary vaccinations plus a booster vaccination at 9-10 months of age. The booster vaccination window was extended up to 18 months of age due to a pause in the study due to the COVID-19 pandemic; actual mean age of booster administration was 12.5 months and ranged from 9 to 16 months.
Period: Overall Study
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Started | 220 | 220 | 220
Received First Vaccination | 220 | 220 | 220
Received Second Vaccination | 217 | 213 | 213
Received Booster Vaccination | 208 | 206 | 206
Completed | 203 | 200 | 200
Not Completed | 17 | 20 | 20
Not completed — Met Ineligibility Criteria During the Study | 1 | 1 | 2
Not completed — Parent Requested Withdrawal | 8 | 12 | 9
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Other | 5 | 6 | 7
Not completed — Lost to Follow-up | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pneumosil | Synflorix | Prevenar 13 | Total
Number analyzed (Participants) | 220 | 220 | 220 | 660
Age, Continuous [Mean (Standard Deviation); unit: days] | 47.3 (3.86) | 46.8 (3.96) | 46.7 (3.74) | 46.9 (3.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 108 | 109 | 342
  Male | 95 | 112 | 111 | 318
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African | 220 | 220 | 220 | 660
Ethnicity [Count of Participants; unit: Participants]
  Mandinka | 109 | 118 | 124 | 351
  Wolof | 21 | 17 | 22 | 60
  Fula | 26 | 25 | 25 | 76
  Jola | 28 | 31 | 15 | 74
  Serahule | 9 | 9 | 9 | 27
  Serere | 9 | 8 | 8 | 25
  Manjago | 5 | 1 | 4 | 10
  Other | 13 | 11 | 13 | 37
Primary Cooking Fuel Source [Count of Participants; unit: Participants]
  Wood/charcoal | 218 | 219 | 219 | 656
  Gas/electricity | 2 | 1 | 1 | 4
Primary Water Source for Cooking/Drinking [Count of Participants; unit: Participants]
  Private tap, well or borehole | 168 | 180 | 178 | 526
  Community tap, well or borehole | 52 | 40 | 42 | 134
Weight [Mean (Standard Deviation); unit: kg] | 4.64 (0.55) | 4.68 (0.58) | 4.67 (0.65) | 4.66 (0.59)
Length [Mean (Standard Deviation); unit: cm] | 55.44 (1.91) | 55.48 (2.02) | 55.29 (2.11) | 55.40 (2.02)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentration (GMC) of Serotype-specific Immunoglobulin G (IgG) Antibodies Four Weeks Post-Booster
Description: The IgG antibody concentration to each of the 10 serotypes contained in Pneumosil was measured by enzyme-linked immunosorbent assay (ELISA) in serum samples collected 4 weeks after the booster dose (Visit 6).
  The pneumococcal serotype-specific IgG ELISAs were performed using the World Health Organisation (WHO) reference assay at the WHO Pneumococcal Serology Reference Laboratory, at the Institute of Child Health, University College London, United Kingdom (UK), where the assay was validated.
Time Frame: 4 weeks post booster dose
Population: Primary Per Protocol Immunogenicity Population (PP_IMM) includes all randomized participants who received all 3 study vaccinations (including booster), contributed post-booster immunogenicity measurements, and with no major protocol deviations that were determined to potentially interfere with immunogenicity assessment. Participants with available data for each serotype are included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 202 | 200 | 200
μg/mL
  Serotype 1: number analyzed (Participants) | 201 | 197 | 200
  Serotype 1 | 8.45 [7.54 to 9.48] | 2.90 [2.57 to 3.28] | 5.87 [5.26 to 6.56]
  Serotype 5: number analyzed (Participants) | 202 | 199 | 200
  Serotype 5 | 1.54 [1.38 to 1.73] | 0.80 [0.72 to 0.88] | 2.04 [1.86 to 2.24]
  Serotype 6A: number analyzed (Participants) | 201 | 195 | 199
  Serotype 6A | 9.56 [8.26 to 11.05] | 0.60 [0.50 to 0.71] | 10.95 [9.57 to 12.54]
  Serotype 6B | 12.46 [11.07 to 14.01] | 4.96 [4.44 to 5.53] | 15.54 [13.71 to 17.60]
  Serotype 7F | 6.66 [5.96 to 7.44] | 3.15 [2.87 to 3.45] | 6.31 [5.75 to 6.93]
  Serotype 9V | 3.46 [3.08 to 3.88] | 2.45 [2.21 to 2.72] | 3.87 [3.47 to 4.32]
  Serotype 14 | 8.28 [6.97 to 9.82] | 5.02 [4.22 to 5.97] | 9.17 [8.06 to 10.45]
  Serotype 19A: number analyzed (Participants) | 200 | 199 | 199
  Serotype 19A | 8.82 [7.65 to 10.15] | 2.39 [1.97 to 2.89] | 12.21 [10.83 to 13.76]
  Serotype 19F: number analyzed (Participants) | 200 | 194 | 197
  Serotype 19F | 11.11 [9.70 to 12.73] | 17.31 [14.83 to 20.20] | 14.99 [13.25 to 16.96]
  Serotype 23F: number analyzed (Participants) | 202 | 200 | 198
  Serotype 23F | 4.95 [4.28 to 5.73] | 2.16 [1.92 to 2.44] | 4.97 [4.34 to 5.69]
Statistical Analysis 1: Comparison: Pneumosil vs Synflorix; Serotype 1 geometric mean concentration ratio (Pneumosil / Synflorix) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 2.91, 95% CI 2-sided [2.47 to 3.44]
Statistical Analysis 2: Comparison: Pneumosil vs Prevenar 13; Serotype 1 geometric mean concentration ratio (Pneumosil / Prevenar 13) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 1.44, 95% CI 2-sided [1.23 to 1.69]
Statistical Analysis 3: Comparison: Pneumosil vs Synflorix; Serotype 5 geometric mean concentration ratio (Pneumosil / Synflorix) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 1.93, 95% CI 2-sided [1.66 to 2.25]
Statistical Analysis 4: Comparison: Pneumosil vs Prevenar 13; Serotype 5 geometric mean concentration ratio (Pneumosil / Prevenar 13) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 0.76, 95% CI 2-sided [0.65 to 0.88]
Statistical Analysis 5: Comparison: Pneumosil vs Synflorix; Serotype 6A geometric mean concentration ratio (Pneumosil / Synflorix) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 16.03, 95% CI 2-sided [12.84 to 20.03]
Statistical Analysis 6: Comparison: Pneumosil vs Prevenar 13; Serotype 6A geometric mean concentration ratio (Pneumosil / Prevenar 13) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 0.87, 95% CI 2-sided [0.72 to 1.06]
Statistical Analysis 7: Comparison: Pneumosil vs Synflorix; Serotype 6B geometric mean concentration ratio (Pneumosil / Synflorix) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 2.51, 95% CI 2-sided [2.14 to 2.95]
Statistical Analysis 8: Comparison: Pneumosil vs Prevenar 13; Serotype 6B geometric mean concentration ratio (Pneumosil / Prevenar 13) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 0.80, 95% CI 2-sided [0.68 to 0.95]
Statistical Analysis 9: Comparison: Pneumosil vs Synflorix; Serotype 7F geometric mean concentration ratio (Pneumosil / Synflorix) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 2.11, 95% CI 2-sided [1.83 to 2.44]
Statistical Analysis 10: Comparison: Pneumosil vs Prevenar 13; Serotype 7F geometric mean concentration ratio (Pneumosil / Prevenar 13) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 1.05, 95% CI 2-sided [0.91 to 1.22]
Statistical Analysis 11: Comparison: Pneumosil vs Synflorix; Serotype 9V geometric mean concentration ratio (Pneumosil / Synflorix) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 1.41, 95% CI 2-sided [1.21 to 1.65]
Statistical Analysis 12: Comparison: Pneumosil vs Prevenar 13; Serotype 9V geometric mean concentration ratio (Pneumosil / Prevenar 13) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 0.89, 95% CI 2-sided [0.76 to 1.05]
Statistical Analysis 13: Comparison: Pneumosil vs Synflorix; Serotype 14 geometric mean concentration ratio (Pneumosil / Synflorix) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 1.65, 95% CI 2-sided [1.29 to 2.10]
Statistical Analysis 14: Comparison: Pneumosil vs Prevenar 13; Serotype 14 geometric mean concentration ratio (Pneumosil / Prevenar 13) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 0.90, 95% CI 2-sided [0.73 to 1.12]
Statistical Analysis 15: Comparison: Pneumosil vs Synflorix; Serotype 19A geometric mean concentration ratio (Pneumosil / Synflorix) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 3.69, 95% CI 2-sided [2.91 to 4.67]
Statistical Analysis 16: Comparison: Pneumosil vs Prevenar 13; Serotype 19A geometric mean concentration ratio (Pneumosil / Prevenar 13) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 0.72, 95% CI 2-sided [0.60 to 0.87]
Statistical Analysis 17: Comparison: Pneumosil vs Synflorix; Serotype 19F geometric mean concentration ratio (Pneumosil / Synflorix) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 0.64, 95% CI 2-sided [0.52 to 0.79]
Statistical Analysis 18: Comparison: Pneumosil vs Prevenar 13; Serotype 19F geometric mean concentration ratio (Pneumosil / Prevenar 13) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 0.74, 95% CI 2-sided [0.62 to 0.89]
Statistical Analysis 19: Comparison: Pneumosil vs Synflorix; Serotype 23F geometric mean concentration ratio (Pneumosil / Synflorix) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 2.29, 95% CI 2-sided [1.89 to 2.76]
Statistical Analysis 20: Comparison: Pneumosil vs Prevenar 13; Serotype 23F geometric mean concentration ratio (Pneumosil / Prevenar 13) and 95% confidence interval (CI). Differences between groups were considered statistically significant if the 95% CI excludes 1; Test type: Other; GMC Ratio = 1.00, 95% CI 2-sided [0.82 to 1.22]

2. Primary Outcome: Number of Participants With Solicited Local and Systemic Adverse Events (AEs) Through Day 6 Following Any Vaccination
Description: Solicited local reactions included tenderness, erythema/redness and induration/swelling at the study vaccine injection site.
  Solicited systemic reactions included cutaneous rash, fever (based on axillary temperature), irritability, drowsiness, and decreased appetite.
  The severity of all solicited AEs was graded from mild (Grade 1) to potentially life threatening (Grade 4), based on protocol-defined criteria that were derived from Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (Version 2.0, November 2014).
Time Frame: Day 0 to Day 6 after each vaccination
Population: The Safety Analysis Set (Safety Population) included all participants who were randomized, received a study vaccination, and provided post-vaccination safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 220 | 220 | 220
Participants
  Any local reaction | 72 | 84 | 63
  Any local reaction Grade 3 or higher | 0 | 0 | 0
  Tenderness | 70 | 83 | 61
  Erythema/Redness | 1 | 3 | 1
  Induration/Swelling | 3 | 5 | 1
  Any systemic reaction | 160 | 167 | 160
  Any systemic reaction Grade 3 or higher | 3 | 0 | 2
  Fever | 98 | 105 | 108
  Fever Grade 3 or higher | 3 | 0 | 2
  Cutaneous Rash | 16 | 7 | 6
  Cutaneous Rash Grade 3 or higher | 0 | 0 | 0
  Irritability | 105 | 110 | 101
  Irritability Grade 3 or higher | 0 | 0 | 0
  Drowsiness | 12 | 15 | 18
  Drowsiness Grade 3 or higher | 0 | 0 | 0
  Decreased Appetite | 25 | 18 | 28
  Decreased Appetite Grade 3 or higher | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Unsolicited Treatment-emergent Adverse Events (TEAEs)
Description: AEs include any intercurrent illness or injury during the study, clinically significant worsening of a preexisting condition, and any solicited AE that occurred or was ongoing 6 days after study vaccine administration. A TEAE is an event that was not present prior to administration of the study vaccine, or increased in intensity after administration of the study vaccine.
  Unsolicited AEs were graded using the scale below:
  Grade 1: Mild; asymptomatic or mild symptoms; intervention not indicated.
  Grade 2: Moderate; minimal, local, or noninvasive intervention indicated.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling.
  Grade 4: Life-threatening consequences; urgent intervention indicated.
  Grade 5: Death related to AE.
  Related AEs are AEs where the Investigator determined a reasonable causal relationship between the vaccine administered and the AE based on medical judgement.
Time Frame: AEs were collected from first dose at age 6 weeks up to 9 months of age, and then from the date of the booster vaccination through 4 weeks post vaccination; approximately 8.5 months overall.
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 220 | 220 | 220
Participants
  Any treatment-emergent adverse event (TEAE) | 198 | 197 | 189
  Any vaccine-related TEAE | 1 | 2 | 0
  Grade 1 TEAE | 196 | 195 | 186
  Vaccine-related Grade 1 TEAE | 1 | 1 | 0
  Grade 2 TEAE | 22 | 20 | 17
  Vaccine-related Grade 2 TEAE | 0 | 0 | 0
  Grade 3 TEAE | 11 | 10 | 6
  Vaccine-related Grade 3 TEAE | 0 | 1 | 0
  Grade 4 TEAE | 0 | 0 | 0
  Grade 5 TEAE | 1 | 0 | 1
  Vaccine related Grade 5 TEAE | 0 | 0 | 0
  TEAEs leading to study discontinuation | 0 | 0 | 1

4. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE was a specific AE that:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of an existing hospitalization.
  * Resulted in a persistent or significant disability or incapacity.
  * Resulted in a congenital anomaly or birth defect
Time Frame: SAEs were collected from first dose at age 6 weeks up to 4 weeks post booster vaccination, approximately 15.5 months overall.
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 220 | 220 | 220
Participants
  Any serious adverse event | 12 | 10 | 7
  Vaccine-related serious adverse events | 0 | 0 | 0

5. Secondary Outcome: Geometric Mean Titers (GMT) of Serotype-specific Opsonophagocytic Activity (OPA) Four Weeks Post-Booster
Description: The functional activity of the antibody response to the 10 serotypes contained in Pneumosil was determined in serum samples collected 4 weeks after the booster dose in a subset of 50 participants per group. This activity was determined using the 4-fold multiplexed opsonophagocytic assay (MOPA) developed at the University of Alabama at Birmingham, and performed at the WHO Pneumococcal Serology Reference Laboratory, at the Institute of Child Health, University College London, UK, where the assay was validated.
  A higher titer indicates increased antibody-mediated opsonophagocytosis.
Time Frame: 4 weeks post booster dose
Population: Primary Per Protocol Immunogenicity population with available serotype data; OPA assays were conducted on the first 50 samples from each treatment group.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 50 | 50 | 50
titer
  Serotype 1: number analyzed (Participants) | 50 | 50 | 49
  Serotype 1 | 631.29 [467.98 to 851.59] | 282.35 [190.44 to 418.60] | 429.13 [310.99 to 592.14]
  Serotype 5 | 885.98 [662.20 to 1185.37] | 484.66 [361.73 to 649.38] | 703.15 [556.01 to 889.24]
  Serotype 6A: number analyzed (Participants) | 50 | 45 | 50
  Serotype 6A | 3651.54 [2593.53 to 5141.16] | 53.86 [25.10 to 115.56] | 6464.88 [5120.52 to 8162.19]
  Serotype 6B | 3931.21 [2969.79 to 5203.89] | 1294.61 [929.52 to 1803.11] | 6012.88 [4130.89 to 8752.29]
  Serotype 7F | 7053.37 [5904.91 to 8425.18] | 4401.18 [3593.44 to 5390.50] | 8288.88 [6756.83 to 10168.3]
  Serotype 9V: number analyzed (Participants) | 50 | 49 | 50
  Serotype 9V | 1408.68 [1092.33 to 1816.64] | 845.47 [631.39 to 1132.13] | 2464.43 [1957.36 to 3102.85]
  Serotype 14 | 2622.36 [1845.88 to 3725.47] | 1381.52 [883.30 to 2160.74] | 3131.96 [2245.73 to 4367.91]
  Serotype 19A | 1620.76 [1200.51 to 2188.13] | 305.46 [177.87 to 524.57] | 3679.06 [2920.79 to 4634.19]
  Serotype 19F | 1384.38 [937.18 to 2044.98] | 2541.40 [1666.99 to 3874.49] | 2094.57 [1410.71 to 3109.94]
  Serotype 23F | 2998.53 [2272.86 to 3955.89] | 1427.66 [1110.72 to 1835.05] | 5687.60 [3891.57 to 8312.54]

6. Secondary Outcome: Percentage of Participants With Serotype-specific Serum IgG Antibody Concentrations ≥ 0.35 μg/mL Four Weeks Post-Booster
Description: The seroresponse rate was defined as the percentage of infants with serotype-specific IgG antibody concentrations of at least 0.35 μg/mL, which is the reference concentration for assessment of vaccine efficacy against invasive pneumococcal diseases (IPDs).
  The IgG concentration to each of the 10 serotypes contained in Pneumosil was measured by ELISA in serum samples collected 4 weeks after the booster dose.
Time Frame: 4 weeks post booster dose
Population: Primary Per Protocol Immunogenicity population with available serotype data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 202 | 200 | 200
percentage of participants
  Serotype 1: number analyzed (Participants) | 201 | 197 | 200
  Serotype 1 | 100 [98.2 to 100.0] | 100 [98.1 to 100.0] | 99.5 [97.3 to 100.0]
  Serotype 5: number analyzed (Participants) | 202 | 199 | 200
  Serotype 5 | 97.5 [94.3 to 99.2] | 89.9 [84.9 to 93.8] | 99.0 [96.4 to 99.9]
  Serotype 6A: number analyzed (Participants) | 201 | 195 | 199
  Serotype 6A | 98.0 [95.0 to 99.5] | 66.2 [59.1 to 72.8] | 99.0 [96.4 to 99.9]
  Serotype 6B | 100 [98.2 to 100.0] | 99.5 [97.3 to 100.0] | 99.5 [97.3 to 100.0]
  Serotype 7F | 100 [98.2 to 100.0] | 99.5 [97.3 to 100.0] | 100 [98.2 to 100.0]
  Serotype 9V | 99.0 [96.5 to 99.9] | 99.5 [97.3 to 100.0] | 100 [98.2 to 100.0]
  Serotype 14 | 98.5 [95.7 to 99.7] | 97.5 [94.3 to 99.2] | 99.5 [97.3 to 100.0]
  Serotype 19A: number analyzed (Participants) | 200 | 199 | 199
  Serotype 19A | 100 [98.2 to 100.0] | 91.5 [86.7 to 94.9] | 100 [98.2 to 100.0]
  Serotype 19F: number analyzed (Participants) | 200 | 194 | 197
  Serotype 19F | 100 [98.2 to 100.0] | 100 [98.1 to 100.0] | 100 [98.1 to 100.0]
  Serotype 23F: number analyzed (Participants) | 202 | 200 | 198
  Serotype 23F | 98.0 [95.0 to 99.5] | 98.0 [95.0 to 99.5] | 98.5 [95.6 to 99.7]

7. Secondary Outcome: Percentage of Participants With Serotype-specific Serum IgG Antibody Concentrations ≥ 1.0 μg/mL Four Weeks Post-Booster
Description: Seroresponse rate was also defined as the percentage of infants with serotype-specific IgG antibody concentrations of at least 1.0 μg/mL.
  The IgG concentration to each of the 10 serotypes contained in Pneumosil was measured by ELISA in serum samples collected 4 weeks after the booster dose.
Time Frame: 4 weeks post booster dose
Population: Primary Per Protocol Immunogenicity population with available data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 202 | 200 | 200
percentage of participants
  Serotype 1: number analyzed (Participants) | 201 | 197 | 200
  Serotype 1 | 98.5 [95.7 to 99.7] | 88.3 [83.0 to 92.5] | 97.5 [94.3 to 99.2]
  Serotype 5: number analyzed (Participants) | 202 | 199 | 200
  Serotype 5 | 68.6 [61.9 to 75.1] | 37.7 [30.9 to 44.8] | 87.5 [82.1 to 91.7]
  Serotype 6A: number analyzed (Participants) | 201 | 195 | 199
  Serotype 6A | 96.5 [93.0 to 98.6] | 37.9 [31.1 to 45.2] | 98.0 [94.9 to 99.5]
  Serotype 6B | 100 [98.2 to 100.0] | 96.5 [92.9 to 98.6] | 99.5 [97.3 to 100.0]
  Serotype 7F | 98.0 [95.0 to 99.5] | 95.0 [91.0 to 97.6] | 99.5 [97.3 to 100.0]
  Serotype 9V | 94.6 [90.5 to 97.3] | 89.5 [84.4 to 93.4] | 95.5 [91.6 to 97.9]
  Serotype 14 | 95.0 [91.1 to 97.6] | 90.0 [85.0 to 93.8] | 99.0 [96.4 to 99.9]
  Serotype 19A: number analyzed (Participants) | 200 | 199 | 199
  Serotype 19A | 96.0 [92.3 to 98.3] | 77.4 [70.9 to 83.0] | 99.5 [97.2 to 100.0]
  Serotype 19F: number analyzed (Participants) | 200 | 194 | 197
  Serotype 19F | 98.5 [95.7 to 99.7] | 96.9 [93.4 to 98.9] | 99.0 [96.4 to 99.9]
  Serotype 23F: number analyzed (Participants) | 202 | 200 | 198
  Serotype 23F | 94.6 [90.5 to 97.3] | 83.0 [77.1 to 87.9] | 96.0 [92.2 to 98.2]

8. Secondary Outcome: Percentage of Participants With Serotype-specific Serum OPA Titers ≥ 8 Four Weeks Post-Booster
Description: The OPA seroresponse rate was defined as the percentage of infants with an OPA titer of at least 8.
  Opsonophagocytic activity was measured using the 4-fold multiplexed opsonophagocytic assay (MOPA) from serum samples taken 4 weeks after the booster vaccination.
Time Frame: 4 weeks post booster dose
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 50 | 50 | 50
percentage of participants
  Serotype 1: number analyzed (Participants) | 50 | 50 | 49
  Serotype 1 | 100 [92.9 to 100.0] | 96.0 [86.3 to 99.5] | 98.0 [89.2 to 100.0]
  Serotype 5 | 100 [92.9 to 100.0] | 100 [92.9 to 100.0] | 100 [92.9 to 100.0]
  Serotype 6A: number analyzed (Participants) | 50 | 45 | 50
  Serotype 6A | 100 [92.9 to 100.0] | 55.6 [40.0 to 70.4] | 100 [92.9 to 100.0]
  Serotype 6B | 100 [92.9 to 100.0] | 98.0 [89.4 to 100.0] | 98.0 [89.4 to 100.0]
  Serotype 7F | 100 [92.9 to 100.0] | 100 [92.9 to 100.0] | 100 [92.9 to 100.0]
  Serotype 9V: number analyzed (Participants) | 50 | 49 | 50
  Serotype 9V | 100 [92.9 to 100.0] | 100 [92.8 to 100.0] | 100 [92.9 to 100.0]
  Serotype 14 | 100 [92.9 to 100.0] | 96.0 [86.3 to 99.5] | 100 [92.9 to 100.0]
  Serotype 19A | 100 [92.9 to 100.0] | 90.0 [78.2 to 96.7] | 100 [92.9 to 100.0]
  Serotype 19F | 98.0 [89.4 to 100.0] | 98.0 [89.4 to 100.0] | 98.0 [89.4 to 100.0]
  Serotype 23F | 100 [92.9 to 100.0] | 100 [92.9 to 100.0] | 100 [92.9 to 100.0]

9. Secondary Outcome: Percentage of Participants With Serotype-specific Serum IgG Antibody Concentrations ≥ 0.35 μg/mL Four Weeks After Completion of Primary Vaccinations
Description: The seroresponse rate was defined as the percentage of infants with serotype-specific IgG antibody concentrations of at least 0.35 μg/mL, which is the reference concentration for assessment of vaccine efficacy against invasive pneumococcal diseases (IPDs).
  The IgG concentration to each of the 10 serotypes contained in Pneumosil was measured by ELISA in serum samples collected 4 weeks after the second primary vaccination dose.
Time Frame: 4 weeks after completion of primary vaccinations (at age 18 weeks)
Population: Primary Per Protocol Immunogenicity population with available serotype data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pneumosil: Infants received two primary vaccinations with Pneumosil, the first at age 6 weeks and the second at age 14 weeks.
- Synflorix: Infants received two primary vaccinations with Synflorix, the first at age 6 weeks and the second at age 14 weeks.
- Prevenar 13: Infants received two primary vaccinations with Prevenar 13, the first at age 6 weeks and the second at age 14 weeks.
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 216 | 212 | 212
percentage of participants
  Serotype 1 | 99.5 [97.5 to 100.0] | 96.2 [92.7 to 98.4] | 100 [98.3 to 100.0]
  Serotype 5 | 96.8 [93.4 to 98.7] | 92.0 [87.5 to 95.3] | 96.2 [92.7 to 98.4]
  Serotype 6A: number analyzed (Participants) | 216 | 211 | 212
  Serotype 6A | 83.3 [77.7 to 88.1] | 12.8 [8.6 to 18.1] | 91.5 [86.9 to 94.9]
  Serotype 6B: number analyzed (Participants) | 216 | 212 | 210
  Serotype 6B | 84.7 [79.2 to 89.2] | 71.2 [64.6 to 77.2] | 89.0 [84.0 to 92.9]
  Serotype 7F | 99.5 [97.5 to 100.0] | 97.2 [93.9 to 99.0] | 100 [98.3 to 100.0]
  Seroytpe 9V | 94.9 [91.1 to 97.4] | 91.0 [86.4 to 94.5] | 98.1 [95.2 to 99.5]
  Serotype 14 | 98.6 [96.0 to 99.7] | 95.3 [91.5 to 97.7] | 97.2 [93.9 to 99.0]
  Serotype 19A: number analyzed (Participants) | 216 | 210 | 212
  Serotype 19A | 97.7 [94.7 to 99.2] | 75.2 [68.8 to 80.9] | 97.6 [94.6 to 99.2]
  Serotype 19F: number analyzed (Participants) | 216 | 209 | 211
  Serotype 19F | 100 [98.3 to 100.0] | 99.5 [97.4 to 100.0] | 100 [98.3 to 100.0]
  Serotype 23F | 95.8 [92.2 to 98.1] | 63.2 [56.3 to 69.7] | 89.6 [84.7 to 93.4]

10. Secondary Outcome: Geometric Mean Concentration of Serotype-specific IgG Antibodies Four Weeks After Completion of Primary Vaccinations
Description: The IgG antibody concentration to each of the 10 serotypes contained in Pneumosil was measured by ELISA in serum samples collected 4 weeks after the second primary vaccination dose.
Time Frame: 4 weeks after completion of primary vaccinations (at age 18 weeks)
Population: Primary Per Protocol Immunogenicity Population with available serotype data
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 216 | 212 | 212
μg/mL
  Serotype 1 | 3.63 [3.32 to 3.98] | 1.36 [1.23 to 1.51] | 3.40 [3.10 to 3.74]
  Serotype 5 | 1.19 [1.10 to 1.28] | 0.87 [0.79 to 0.96] | 1.81 [1.62 to 2.01]
  Serotype 6A: number analyzed (Participants) | 216 | 211 | 212
  Serotype 6A | 1.19 [1.00 to 1.41] | 0.14 [0.13 to 0.16] | 2.62 [2.24 to 3.08]
  Serotype 6B: number analyzed (Participants) | 216 | 212 | 210
  Serotype 6B | 1.82 [1.48 to 2.23] | 0.91 [0.75 to 1.10] | 1.75 [1.49 to 2.07]
  Serotype 7F | 3.46 [3.09 to 3.88] | 1.73 [1.55 to 1.92] | 4.67 [4.19 to 5.20]
  Serotype 9V | 1.93 [1.74 to 2.16] | 1.31 [1.17 to 1.46] | 2.56 [2.28 to 2.88]
  Serotype 14 | 4.03 [3.50 to 4.64] | 2.58 [2.18 to 3.04] | 3.27 [2.70 to 3.96]
  Serotype 19A: number analyzed (Participants) | 216 | 210 | 212
  Serotype 19A | 1.75 [1.57 to 1.96] | 0.65 [0.57 to 0.73] | 4.38 [3.73 to 5.15]
  Serotype 19F: number analyzed (Participants) | 216 | 209 | 211
  Serotype 19F | 5.45 [4.94 to 6.01] | 8.86 [7.71 to 10.17] | 9.06 [7.97 to 10.30]
  Serotype 23F | 2.21 [1.92 to 2.56] | 0.57 [0.48 to 0.68] | 1.64 [1.39 to 1.93]

11. Secondary Outcome: Percentage of Participants With Serotype-specific Serum OPA Titers ≥ 8 Four Weeks After Completion of Primary Vaccinations
Description: The OPA seroresponse rate was defined as the percentage of infants with an OPA titer of at least 8.
  Opsonophagocytic activity was measured using the 4-fold multiplexed opsonophagocytic assay (MOPA).
Time Frame: 4 weeks after completion of primary vaccinations (at age 18 weeks)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 50 | 50 | 50
percentage of participants
  Serotype 1: number analyzed (Participants) | 50 | 49 | 50
  Serotype 1 | 98.0 [89.4 to 100.0] | 73.5 [58.9 to 85.1] | 96.0 [86.3 to 99.5]
  Serotype 5 | 98.0 [89.4 to 100.0] | 96.0 [86.3 to 99.5] | 100 [92.9 to 100.0]
  Serotype 6A: number analyzed (Participants) | 50 | 49 | 50
  Serotype 6A | 92.0 [80.8 to 97.8] | 10.2 [3.4 to 22.2] | 98.0 [89.4 to 100.0]
  Serotype 6B: number analyzed (Participants) | 50 | 49 | 50
  Serotype 6B | 96.0 [86.3 to 99.5] | 69.4 [54.6 to 81.8] | 92.0 [80.8 to 97.8]
  Serotype 7F | 100 [92.9 to 100.0] | 100 [92.9 to 100.0] | 100 [92.9 to 100.0]
  Serotype 9V: number analyzed (Participants) | 47 | 50 | 50
  Serotype 9V | 100 [92.5 to 100.0] | 100 [92.9 to 100.0] | 100 [92.9 to 100.0]
  Serotype 14: number analyzed (Participants) | 50 | 48 | 50
  Serotype 14 | 94.0 [83.5 to 98.8] | 97.9 [88.9 to 100.0] | 90.0 [78.2 to 96.7]
  Serotype 19A: number analyzed (Participants) | 49 | 46 | 50
  Serotype 19A | 91.8 [80.4 to 97.7] | 56.5 [41.1 to 71.1] | 96.0 [86.3 to 99.5]
  Serotype 19F: number analyzed (Participants) | 50 | 49 | 50
  Serotype 19F | 96.0 [86.3 to 99.5] | 95.9 [86.0 to 99.5] | 98.0 [89.4 to 100.0]
  Serotype 23F: number analyzed (Participants) | 48 | 47 | 49
  Serotype 23F | 100 [92.6 to 100.0] | 100 [92.5 to 100.0] | 100 [92.8 to 100.0]

12. Secondary Outcome: Geometric Mean Titers of Serotype-specific Serum OPA Four Weeks After Primary Vaccinations
Description: Opsonophagocytic activity was measured using the 4-fold multiplexed opsonophagocytic assay (MOPA).
Time Frame: 4 weeks after completion of primary vaccinations (at age 18 weeks)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 50 | 50 | 50
titer
  Serotype 1: number analyzed (Participants) | 50 | 49 | 50
  Serotype 1 | 99.67 [71.83 to 138.30] | 26.70 [17.72 to 40.22] | 98.63 [70.61 to 137.78]
  Serotype 5 | 182.18 [134.53 to 246.70] | 85.09 [58.98 to 122.75] | 291.98 [221.91 to 384.18]
  Serotype 6A: number analyzed (Participants) | 50 | 49 | 50
  Serotype 6A | 400.49 [238.40 to 672.79] | 5.35 [4.04 to 7.08] | 1524.31 [1066.28 to 2179.09]
  Serotype 6B: number analyzed (Participants) | 50 | 49 | 50
  Serotype 6B | 923.86 [589.56 to 1447.73] | 166.74 [88.71 to 313.43] | 920.43 [573.35 to 1477.61]
  Serotype 7F | 2069.84 [1622.83 to 2639.98] | 1096.84 [853.88 to 1408.93] | 3069.95 [2435.98 to 3868.91]
  Serotype 9V: number analyzed (Participants) | 47 | 50 | 50
  Serotype 9V | 134.50 [87.35 to 207.10] | 58.24 [38.29 to 88.58] | 331.79 [241.48 to 455.89]
  Serotype 14: number analyzed (Participants) | 50 | 48 | 50
  Serotype 14 | 669.79 [383.93 to 1168.50] | 577.98 [376.06 to 888.33] | 489.56 [224.00 to 1069.94]
  Serotype 19A: number analyzed (Participants) | 49 | 46 | 50
  Serotype 19A | 69.15 [46.95 to 101.85] | 22.40 [13.27 to 37.83] | 324.64 [204.39 to 515.65]
  Serotype 19F: number analyzed (Participants) | 50 | 49 | 50
  Serotype 19F | 381.46 [269.27 to 540.40] | 690.36 [461.10 to 1033.61] | 647.79 [460.50 to 911.24]
  Serotype 23F: number analyzed (Participants) | 48 | 47 | 49
  Serotype 23F | 806.12 [584.18 to 1112.39] | 180.97 [106.19 to 308.44] | 748.96 [458.35 to 1223.84]

13. Secondary Outcome: Percentage of Participants With Serotype-specific Serum IgG Concentrations ≥ 0.35 μg/mL Prior to Booster
Description: The seroresponse rate was defined as the percentage of infants with serotype-specific IgG concentrations of at least 0.35 μg/mL, which is the reference concentration for assessment of vaccine efficacy against invasive pneumococcal diseases (IPDs).
  The IgG concentration to each of the 10 serotypes contained in Pneumosil was measured by ELISA in serum samples collected immediately prior to the booster vaccination dose.
Time Frame: Prior to the booster dose at approximately 9 to 16 months of age
Population: Primary Per Protocol Immunogenicity population with available serotype data
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 208 | 206 | 206
percentage of participants
  Serotype 1: number analyzed (Participants) | 207 | 203 | 206
  Serotype 1 | 50.2 [43.2 to 57.3] | 17.2 [12.3 to 23.2] | 53.4 [46.3 to 60.4]
  Serotype 5: number analyzed (Participants) | 205 | 201 | 204
  Serotype 5 | 13.7 [9.3 to 19.1] | 16.4 [11.6 to 22.3] | 33.8 [27.4 to 40.8]
  Serotype 6A: number analyzed (Participants) | 208 | 205 | 206
  Serotype 6A | 76.0 [69.6 to 81.6] | 32.7 [26.3 to 39.6] | 70.4 [63.7 to 76.5]
  Serotype 6B: number analyzed (Participants) | 208 | 205 | 206
  Serotype 6B | 89.9 [85.0 to 93.6] | 74.6 [68.1 to 80.4] | 60.7 [53.7 to 67.4]
  Serotype 7F: number analyzed (Participants) | 208 | 205 | 206
  Serotype 7F | 74.5 [68.0 to 80.3] | 65.4 [58.4 to 71.9] | 84.5 [78.8 to 89.1]
  Serotype 9V: number analyzed (Participants) | 205 | 205 | 204
  Serotype 9V | 35.1 [28.6 to 42.1] | 36.1 [29.5 to 43.1] | 37.7 [31.1 to 44.8]
  Serotype 14: number analyzed (Participants) | 207 | 204 | 205
  Serotype 14 | 69.6 [62.8 to 75.8] | 59.3 [52.2 to 66.1] | 86.3 [80.9 to 90.7]
  Serotype 19A: number analyzed (Participants) | 203 | 204 | 204
  Serotype 19A | 58.1 [51.0 to 65.0] | 54.9 [47.8 to 61.9] | 65.7 [58.7 to 72.2]
  Serotype 19F: number analyzed (Participants) | 207 | 205 | 206
  Serotype 19F | 84.1 [78.4 to 88.8] | 95.1 [91.2 to 97.6] | 80.6 [74.5 to 85.8]
  Serotype 23F: number analyzed (Participants) | 208 | 206 | 205
  Serotype 23F | 46.2 [39.2 to 53.2] | 19.4 [14.3 to 25.5] | 24.9 [19.1 to 31.4]

14. Secondary Outcome: Geometric Mean Concentration of Serotype-specific Serum IgG Antibodies Prior to Booster
Description: The IgG antibody concentration to each of the 10 serotypes contained in Pneumosil was measured by ELISA in serum samples collected immediately prior to the booster vaccination dose.
Time Frame: Prior to the booster dose at approximately 9 to 16 months of age
Population: Primary Per Protocol Immunogenicity population with available serotype data
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 208 | 206 | 206
μg/mL
  Serotype 1: number analyzed (Participants) | 207 | 203 | 206
  Serotype 1 | 0.36 [0.33 to 0.41] | 0.16 [0.15 to 0.18] | 0.37 [0.33 to 0.41]
  Serotype 5: number analyzed (Participants) | 205 | 201 | 204
  Serotype 5 | 0.17 [0.15 to 0.18] | 0.16 [0.14 to 0.17] | 0.24 [0.22 to 0.27]
  Serotype 6A: number analyzed (Participants) | 208 | 205 | 206
  Serotype 6A | 0.62 [0.55 to 0.70] | 0.22 [0.19 to 0.25] | 0.50 [0.45 to 0.56]
  Serotype 6B: number analyzed (Participants) | 208 | 205 | 206
  Serotype 6B | 0.97 [0.87 to 1.08] | 0.56 [0.50 to 0.62] | 0.45 [0.39 to 0.50]
  Serotype 7F: number analyzed (Participants) | 208 | 205 | 206
  Serotype 7F | 0.60 [0.53 to 0.68] | 0.43 [0.39 to 0.48] | 0.72 [0.64 to 0.80]
  Serotype 9V: number analyzed (Participants) | 205 | 205 | 204
  Serotype 9V | 0.25 [0.23 to 0.28] | 0.29 [0.26 to 0.32] | 0.28 [0.25 to 0.31]
  Serotype 14: number analyzed (Participants) | 207 | 204 | 205
  Serotype 14 | 0.71 [0.60 to 0.83] | 0.48 [0.41 to 0.56] | 1.16 [1.00 to 1.35]
  Serotype 19A: number analyzed (Participants) | 203 | 204 | 204
  Serotype 19A | 0.49 [0.42 to 0.56] | 0.40 [0.35 to 0.45] | 0.53 [0.46 to 0.62]
  Serotype 19F: number analyzed (Participants) | 207 | 205 | 206
  Serotype 19F | 0.83 [0.73 to 0.94] | 1.25 [1.11 to 1.40] | 0.72 [0.63 to 0.83]
  Serotype 23F: number analyzed (Participants) | 208 | 206 | 205
  Serotype 23F | 0.32 [0.27 to 0.37] | 0.16 [0.15 to 0.19] | 0.17 [0.15 to 0.20]

15. Secondary Outcome: Percentage of Participants With Serotype-specific Serum OPA Titers ≥ 8 Prior to Booster
Description: The OPA seroresponse rate was defined as the percentage of infants with an OPA titer of at least 8.
  Opsonophagocytic activity was measured using the 4-fold multiplexed opsonophagocytic assay (MOPA) from serum samples collected immediately prior to the booster vaccination dose.
Time Frame: Prior to the booster dose at approximately 9 to 16 months of age
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 50 | 50 | 50
percentage of participants
  Serotype 1: number analyzed (Participants) | 49 | 50 | 47
  Serotype 1 | 22.4 [11.8 to 36.6] | 16.0 [7.2 to 29.1] | 25.5 [13.9 to 40.3]
  Serotype 5: number analyzed (Participants) | 48 | 49 | 49
  Serotype 5 | 58.3 [43.2 to 72.4] | 49.0 [34.4 to 63.7] | 63.3 [48.3 to 76.6]
  Serotype 6A: number analyzed (Participants) | 47 | 50 | 47
  Serotype 6A | 76.6 [62.0 to 87.7] | 14.0 [5.8 to 26.7] | 63.8 [48.5 to 77.3]
  Serotype 6B: number analyzed (Participants) | 48 | 48 | 48
  Serotype 6B | 87.5 [74.8 to 95.3] | 62.5 [47.3 to 76.1] | 54.2 [39.2 to 68.6]
  Serotype 7F: number analyzed (Participants) | 49 | 49 | 48
  Serotype 7F | 100 [92.8 to 100.0] | 100 [92.8 to 100.0] | 100 [92.6 to 100.0]
  Serotype 9V: number analyzed (Participants) | 44 | 43 | 45
  Serotype 9V | 100 [92.0 to 100.0] | 100 [91.8 to 100.0] | 100 [92.1 to 100.0]
  Serotype 14: number analyzed (Participants) | 49 | 48 | 48
  Serotype 14 | 75.5 [61.1 to 86.7] | 52.1 [37.2 to 66.7] | 72.9 [58.2 to 84.7]
  Serotype 19A: number analyzed (Participants) | 48 | 49 | 49
  Serotype 19A | 35.4 [22.2 to 50.5] | 40.8 [27.0 to 55.8] | 63.3 [48.3 to 76.6]
  Serotype 19F: number analyzed (Participants) | 48 | 49 | 49
  Serotype 19F | 60.4 [45.3 to 74.2] | 79.6 [65.7 to 89.8] | 36.7 [23.4 to 51.7]
  Serotype 23F: number analyzed (Participants) | 43 | 42 | 42
  Serotype 23F | 100 [91.8 to 100.0] | 100 [91.6 to 100.0] | 100 [91.6 to 100.0]

16. Secondary Outcome: Geometric Mean Titer of Serotype-specific Serum OPA Prior to Booster
Description: Opsonophagocytic activity was measured using the 4-fold multiplexed opsonophagocytic assay (MOPA) from serum samples collected immediately prior to the booster vaccination dose.
Time Frame: Prior to the booster dose at approximately 9 to 16 months of age
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 50 | 50 | 50
titer
  Serotype 1: number analyzed (Participants) | 49 | 50 | 47
  Serotype 1 | 5.57 [4.56 to 6.80] | 5.19 [4.27 to 6.30] | 5.45 [4.57 to 6.49]
  Serotype 5: number analyzed (Participants) | 48 | 49 | 49
  Serotype 5 | 12.53 [9.03 to 17.37] | 12.01 [8.28 to 17.43] | 16.03 [10.95 to 23.45]
  Serotype 6A: number analyzed (Participants) | 47 | 50 | 47
  Serotype 6A | 42.59 [26.46 to 68.55] | 6.41 [4.49 to 9.15] | 40.66 [22.34 to 74.00]
  Serotype 6B: number analyzed (Participants) | 48 | 48 | 48
  Serotype 6B | 121.60 [78.09 to 189.36] | 40.08 [25.20 to 63.72] | 32.27 [19.77 to 52.68]
  Serotype 7F: number analyzed (Participants) | 49 | 49 | 48
  Serotype 7F | 1756.80 [1234.91 to 2499.24] | 1725.63 [1206.66 to 2467.79] | 1688.30 [1160.23 to 2456.74]
  Serotype 9V: number analyzed (Participants) | 44 | 43 | 45
  Serotype 9V | 27.60 [15.80 to 48.21] | 27.95 [17.48 to 44.67] | 48.64 [29.08 to 81.36]
  Serotype 14: number analyzed (Participants) | 49 | 48 | 48
  Serotype 14 | 60.53 [32.55 to 112.55] | 17.67 [10.31 to 30.29] | 62.77 [33.95 to 116.08]
  Serotype 19A: number analyzed (Participants) | 48 | 49 | 49
  Serotype 19A | 13.43 [7.80 to 23.11] | 12.88 [8.25 to 20.12] | 28.20 [16.96 to 46.89]
  Serotype 19F: number analyzed (Participants) | 48 | 49 | 49
  Serotype 19F | 24.09 [13.90 to 41.77] | 57.66 [33.74 to 98.52] | 12.27 [7.34 to 20.50]
  Serotype 23F: number analyzed (Participants) | 43 | 42 | 42
  Serotype 23F | 65.62 [38.19 to 112.74] | 41.99 [23.29 to 75.68] | 81.42 [44.08 to 150.40]

17. Secondary Outcome: Ratio of Serotype-specific Serum IgG GMC 4 Weeks Post-Booster to Serotype-specific IgG GMC 4 Weeks After Completion of Primary Vaccinations
Description: Booster response was measured by the ratio of IgG GMCs measured at the post-booster visit to those measured 4 weeks after completion of primary vaccinations.
Time Frame: 4 weeks after completion of primary vaccinations (at age 18 weeks) and 4 weeks post booster
Population: Primary Per Protocol Immunogenicity population with available data for each serotype at both time points
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 202 | 200 | 200
ratio
  Serotype 1: number analyzed (Participants) | 201 | 197 | 200
  Serotype 1 | 2.31 [2.10 to 2.55] | 2.09 [1.86 to 2.34] | 1.74 [1.54 to 1.97]
  Serotype 5: number analyzed (Participants) | 202 | 199 | 200
  Serotype 5 | 1.29 [1.15 to 1.44] | 0.90 [0.81 to 1.01] | 1.15 [1.02 to 1.30]
  Serotype 6A: number analyzed (Participants) | 201 | 195 | 199
  Serotype 6A | 7.86 [6.54 to 9.44] | 4.30 [3.61 to 5.12] | 4.14 [3.49 to 4.91]
  Serotype 6B: number analyzed (Participants) | 202 | 200 | 198
  Serotype 6B | 6.71 [5.48 to 8.21] | 5.32 [4.46 to 6.35] | 8.92 [7.47 to 10.66]
  Serotype 7F | 1.91 [1.69 to 2.17] | 1.84 [1.64 to 2.05] | 1.36 [1.22 to 1.52]
  Serotype 9V | 1.76 [1.55 to 1.98] | 1.86 [1.65 to 2.09] | 1.55 [1.34 to 1.79]
  Serotype 14 | 1.98 [1.69 to 2.33] | 1.93 [1.61 to 2.33] | 2.80 [2.29 to 3.43]
  Serotype 19A: number analyzed (Participants) | 200 | 197 | 199
  Serotype 19A | 4.98 [4.33 to 5.74] | 3.69 [3.08 to 4.42] | 2.69 [2.25 to 3.22]
  Serotype 19F: number analyzed (Participants) | 200 | 192 | 196
  Serotype 19F | 1.98 [1.74 to 2.26] | 1.96 [1.68 to 2.29] | 1.68 [1.46 to 1.94]
  Serotype 23F: number analyzed (Participants) | 202 | 200 | 198
  Serotype 23F | 2.24 [1.95 to 2.58] | 3.67 [3.10 to 4.36] | 3.00 [2.55 to 3.52]

18. Secondary Outcome: Ratio of Serotype-specific Serum OPA GMT 4 Weeks Post-Booster to Serotype-specific OPA GMT 4 Weeks After Completion of Primary Vaccinations
Description: OPA booster response was measured by the ratio of OPA GMTs measured at the post-booster visit to those measured 4 weeks after completion of primary vaccinations.
Time Frame: 4 weeks after completion of primary vaccinations (at age 18 weeks) and 4 weeks post booster
Population: Primary Per Protocol Immunogenicity population with available data for each serotype at both time points; OPA assays were conducted on the first 50 samples from each treatment group.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Pneumosil | Synflorix | Prevenar 13
Number analyzed (Participants) | 50 | 50 | 50
ratio
  Serotype 1: number analyzed (Participants) | 50 | 49 | 49
  Serotype 1 | 6.70 [5.07 to 8.86] | 9.35 [6.50 to 13.46] | 4.45 [2.94 to 6.74]
  Serotype 5 | 4.91 [3.71 to 6.49] | 5.36 [3.78 to 7.61] | 2.46 [1.86 to 3.25]
  Serotype 6A: number analyzed (Participants) | 50 | 45 | 50
  Serotype 6A | 10.36 [6.54 to 16.41] | 10.12 [4.98 to 20.53] | 3.89 [2.70 to 5.61]
  Serotype 6B: number analyzed (Participants) | 50 | 49 | 50
  Serotype 6B | 4.62 [2.84 to 7.53] | 7.70 [4.40 to 13.46] | 6.54 [4.03 to 10.60]
  Serotype 7F | 3.51 [2.67 to 4.62] | 4.03 [2.93 to 5.54] | 2.71 [2.08 to 3.53]
  Serotype 9V: number analyzed (Participants) | 47 | 49 | 50
  Serotype 9V | 10.24 [6.36 to 16.50] | 14.90 [9.12 to 24.35] | 7.64 [5.58 to 10.45]
  Serotype 14: number analyzed (Participants) | 50 | 48 | 50
  Serotype 14 | 4.27 [2.38 to 7.64] | 2.25 [1.32 to 3.83] | 5.73 [2.84 to 11.60]
  Serotype 19A: number analyzed (Participants) | 49 | 46 | 50
  Serotype 19A | 23.79 [15.61 to 36.25] | 12.25 [6.86 to 21.87] | 11.63 [7.59 to 17.81]
  Serotype 19F: number analyzed (Participants) | 50 | 49 | 50
  Serotype 19F | 3.74 [2.47 to 5.65] | 3.30 [2.32 to 4.68] | 3.55 [2.35 to 5.39]
  Serotype 23F: number analyzed (Participants) | 48 | 47 | 49
  Serotype 23F | 3.81 [2.69 to 5.40] | 8.71 [5.63 to 13.45] | 7.41 [4.32 to 12.72]

ADVERSE EVENTS:
Time Frame: All-cause mortality and SAEs were collected from first dose at age 6 weeks up to 4 weeks post booster vaccination, approximately 15.5 months overall. Non-serious AEs were collected from first dose at age 6 weeks up to 9 months of age, and then from the date of the booster vaccination through 4 weeks post booster vaccination; approximately 8.5 months overall.
Description: Data reported Include both solicited and unsolicited events.
Arm/Group | Pneumosil | Synflorix | Prevenar 13
All-Cause Mortality (participants affected / at risk) | 1/220 | 0/220 | 1/220
Serious Adverse Events (participants affected / at risk) | 12/220 | 10/220 | 7/220
Other Adverse Events (participants affected / at risk) | 212/220 | 213/220 | 211/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pneumosil (N=220) | Synflorix (N=220) | Prevenar 13 (N=220)
Gastroenteritis (Infections and infestations) | 5 | 2 | 0
Bronchiolitis (Infections and infestations) | 3 | 1 | 2
Periorbital cellulitis (Infections and infestations) | 0 | 3 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2 | 1
Infected dermal cyst (Infections and infestations) | 0 | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0
Vulval cellulitis (Infections and infestations) | 1 | 0 | 0
Atrioventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1 | 0
Sickle cell anaemia (Congenital, familial and genetic disorders) | 1 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pneumosil (N=220) | Synflorix (N=220) | Prevenar 13 (N=220)
Upper respiratory tract infection (Infections and infestations) | 111 | 112 | 99
Furuncle (Infections and infestations) | 52 | 40 | 39
Conjunctivitis (Infections and infestations) | 29 | 42 | 36
Gastroenteritis (Infections and infestations) | 24 | 21 | 29
Rash pustular (Infections and infestations) | 18 | 16 | 22
Skin candida (Infections and infestations) | 22 | 11 | 17
Body tinea (Infections and infestations) | 13 | 12 | 14
Pneumonia (Infections and infestations) | 11 | 10 | 17
Bronchiolitis (Infections and infestations) | 10 | 8 | 12
Otitis media (Infections and infestations) | 8 | 8 | 9
Febrile infection (Infections and infestations) | 7 | 8 | 9
Impetigo (Infections and infestations) | 9 | 11 | 7
Oral candidiasis (Infections and infestations) | 6 | 7 | 5
Tinea capitis (Infections and infestations) | 6 | 6 | 4
Tinea infection (Infections and infestations) | 7 | 1 | 7
Cutaneous larva migrans (Infections and infestations) | 6 | 1 | 7
Abscess (Infections and infestations) | 2 | 5 | 2
Otitis media acute (Infections and infestations) | 3 | 5 | 1
Nasopharyngitis (Infections and infestations) | 4 | 1 | 1
Tinea versicolour (Infections and infestations) | 1 | 4 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 3
Abscess limb (Infections and infestations) | 1 | 2 | 1
Otitis externa (Infections and infestations) | 1 | 1 | 2
Varicella (Infections and infestations) | 3 | 1 | 0
Pustule (Infections and infestations) | 1 | 1 | 1
Vaccination site abscess (Infections and infestations) | 1 | 1 | 1
Acarodermatitis (Infections and infestations) | 1 | 0 | 1
Dysentery (Infections and infestations) | 1 | 1 | 0
Infected dermal cyst (Infections and infestations) | 0 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 1
Viral rash (Infections and infestations) | 0 | 1 | 1
Angular cheilitis (Infections and infestations) | 0 | 1 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 1
Candida nappy rash (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Dermatophytosis (Infections and infestations) | 0 | 0 | 1
Gingival abscess (Infections and infestations) | 0 | 1 | 0
Helminthic infection (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0
Mastitis (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Vaccination site infection (Infections and infestations) | 1 | 0 | 0
Vaccination site pustule (Infections and infestations) | 0 | 1 | 0
Irritability postvaccinal (General disorders) | 105 | 110 | 101
Pyrexia (General disorders) | 96 | 104 | 108
Vaccination site pain (General disorders) | 70 | 83 | 61
Vaccination site induration (General disorders) | 3 | 5 | 1
Vaccination site erythema (General disorders) | 1 | 3 | 1
Vaccination site swelling (General disorders) | 1 | 0 | 1
Developmental delay (General disorders) | 0 | 1 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 52 | 58 | 45
Vomiting (Gastrointestinal disorders) | 8 | 9 | 6
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 3 | 2
Infantile colic (Gastrointestinal disorders) | 3 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 25 | 29 | 15
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 14 | 10 | 13
Rash (Skin and subcutaneous tissue disorders) | 12 | 6 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 8 | 4 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 7 | 4 | 2
Rash vesicular (Skin and subcutaneous tissue disorders) | 4 | 5 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Exfoliative rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 25 | 18 | 29
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 1
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 12 | 15 | 18
Infant irritability (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 7 | 7 | 6
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tooth injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 3
Conjunctivitis allergic (Eye disorders) | 4 | 1 | 0
Blepharitis (Eye disorders) | 2 | 1 | 1
Vernal keratoconjunctivitis (Eye disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 2
Pulmonary valve stenosis (Cardiac disorders) | 0 | 0 | 1
Cystic lymphangioma (Congenital, familial and genetic disorders) | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT03896477/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT03896477/SAP_001.pdf